CLINICAL TRIAL: NCT05520697
Title: Effect of a Physical Training Program on Cerebral Hemodynamics in Patients With Metabolic-associated Fatty Liver Disease
Brief Title: Exercise and Cerebral Hemodynamics in MAFLD.
Acronym: CERHEMAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Ricardo U. Macías-Rodríguez, Assistant Professor Hepatology/Clinical Researcher, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAS-3608-21-23-1
Record Dates: First submitted 2022-08-23; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Nutritional treatment with caloric restriction and mental exercise
  Interventions: Behavioral: Nutritional intervention; Behavioral: Mental exercise.
- Intervention (Experimental): Nutritional treatment with caloric restriction, mental exercise, and physical training program.
  Interventions: Behavioral: Nutritional intervention; Behavioral: Mental exercise.; Behavioral: Physical training.

INTERVENTIONS:
Behavioral: Nutritional intervention — Nutritional treatment with caloric restriction.
Behavioral: Mental exercise. — Mental exercise.
Behavioral: Physical training. — Exercise.
  Arms: Intervention

SUMMARY:
Arterial stiffness and endothelial dysfunction present in metabolic associated fatty liver disease (MAFLD) confer increased cardiovascular risk, which represents the leading cause of mortality in this group of patients.

Mechanisms involved in the cardiovascular complications of MAFLD have recently been found to also affect cerebral blood flow altering cerebral hemodynamics in MAFLD subjects. These alerations can be detected through transcranial Doppler, which measures markers of cerebrovascular vasoconstriction, which indicates cerebrovascular autoregulation.16 These abnormalities are related to vascular disease in MAFLD, which plays an essential role in ischemic stroke and cognitive impairment, which explains why MAFLD patients had lower scores on cognitive function tests.17 Nonetheless, there are no studies evaluating the effect of lifestyle interventions (specifically exercise) on cerebral hemodynamics in patients with MAFLD, however, it has been shown that in other pathologies that share pathophysiological similarities with NAFLD there are beneficial changes in this outcome. An example of the above is chronic heart failure and liver cirrhosis, where physical exercise attenuates the inflammatory cascade (decrease in IL6, IL8, IL12, TNFa), and decreases the activation of the renin-angiotensin system with a direct effect on endothelial function improvement. Our research group also documented that a 12-week physical training program acts on this mechanism and has a beneficial effect on cerebral hemodynamics evaluated by transcranial Doppler in patients with liver cirrhosis, which leads to an improvement in neuropsychometric tests.18 Improvement in the previously described pathways through a 16-week physical training program in MAFLD patients could potentially improve alterations in cerebral blood flow, cognitive function, endothelial function, body composition, and the degree of liver steatosis and fibrosis. This outcome has never been assessed in MAFLD patients undergoing exercise. In addition, although there are studies that demonstrate the impact of diet and exercise, most have evaluated these interventions individually, which represents a limitation when implementing them as a multidisciplinary intervention.

Therefore, our hypothesis is that a 16-week physical training program will improve cerebral hemodynamic parameters in patients with metabolic-associated fatty liver compared to a control group without a physical training program.

DETAILED DESCRIPTION:
Hepatic steatosis associated with metabolic dysfunction, abbreviated as MAFLD (Metabolic Associated Fatty Liver Disease) is currently the most common liver disease and has become one of the main etiologies of chronic liver disease and hepatocellular carcinoma (HCC) in the western world, it is estimated that in a few years it will be the leading cause of liver cirrhosis1.

MAFLD encompasses a broad spectrum of liver injury of varying severity ranging from simple steatosis to steatohepatitis (NASH). In principle, simple steatosis is the accumulation of lipids in more than 5% of hepatocytes, but it can progress in approximately 10-20% of subjects with simple steatosis to steatohepatitis which is defined as steatosis accompanied by cell ballooning, lobular inflammation, and fibrosis, and if this persists without treatment, up to 10-25% may progress to liver cirrhosis and/or hepatocellular carcinoma .2,3 Epidemiology MAFLD is a common disease worldwide and presents a significant burden on health systems. It is present in 6-25% of the world population. In Latin America, the prevalence ranges between 17% to 33%, while in Mexico the prevalence is 14-30% in the general population.4 MAFLD is more common in patients in their fifth decade of life, and there are groups at higher risk, such as subjects with Type 2 Diabetes Mellitus (DM2) and patients with dyslipidemia, where the frequency of the disease increases to 62% and 83% respectively.5 Due to the increasing trend of obesity, the incidence rate of NAFLD is expected to increase significantly in the coming decades; in fact, only 3-20% of patients with this pathology are not obese, so it is concluded that obesity is the most common clinical phenotype associated with MAFLD.4,5 MAFLD-associated complications Obesity has been linked not only to simple steatosis but also to advanced disease, i.e., NASH. As a consequence, in addition to increasing all-cause mortality, obesity appears to increase liver-specific mortality in patients with MAFLD, and due to the lack of approved pharmacological interventions to counteract the disease, targeting obesity is considered an option. essential for its management.6 In NAFLD, as in other metabolic disorders, there is low-grade inflammation that is mainly determined by the expansion of visceral adipose tissue, which produces proinflammatory cytokines (IL-1B, IL-6, and TNF-a) that cause both inflammation at the hepatic level through the portal route, as well as systemic inflammation with repercussions in different organs and tissues, including muscle, heart, and brain.7 These characteristics in combination with the release of pro-coagulant, pro-oxidant, and pro-fibrogenic factors represent a risk factor for endothelial dysfunction and vascular damage. Additionally, MAFLD is associated with an increase in components of the renin-angiotensin system, particularly angiotensin II, which may contribute to vascular damage by increasing oxidative stress and accelerating atherosclerosis7,8 The mechanisms described suggest that in MAFLD, vascular alterations and endothelial dysfunction, in addition to the known manifestations of cardiovascular risk, lead to incipient alterations in cerebral blood flow (microvascular) that contribute to cognitive deterioration and increase the risk of ischemic stroke. In fact, MAFLD is associated with ischemic stroke even after adjustment for other cardiovascular risk factors such as obesity, dyslipidemia, and type 2 DM.9,10 Pharmacological and non-pharmacological treatment in MAFLD There is no registered effective pharmacological treatment for MAFLD, but guidelines support the use of vitamin E in MAFLD subjects without type 2 diabetes, or pioglitazone in NASH patients, and four drugs (obeticholic acid, elafibranor, selonsertib, and cenicriviroc) have entered phase III of development.11 Due to the above, lifestyle modification to achieve weight reduction represents the first-line treatment for MAFLD and resolves hepatic steatosis and hepatic fibrosis.12 Loss of at least 7% of body weight is associated with improvement in steatosis, but greater weight loss (>10%) is needed to reverse the histopathologic features of NASH, including fibrosis. In obese subjects a reduction of 1 kg/week is suggested and in morbid obesity 1.5-2.5 kg/week; Weight loss greater than these amounts is associated with adverse effects, such as an increased inflammatory state in these patients, and increased mobilization of intrahepatic fat, which is associated with worsening hepatic steatosis.12 Although nutritional management is the cornerstone of MAFLD treatment, physical activity should always be part of comprehensive management. Exercise intervention studies in MAFLD have shown that both aerobic and resistance exercise significantly decrease intrahepatic lipid content. In addition, there is evidence that exercise has a role in improving endothelial dysfunction in patients with MAFLD, which could have implications for the prevention of cardiovascular diseases. These benefits appear to be independent of exercise intensity and dose.13 The exact mechanisms by which exercise decreases intrahepatic lipid content are not fully understood. Some studies reported that the improvement is related to weight loss, while others reported an independent benefit.14 Several pathways could be involved in this improvement, such as decreasing insulin resistance, modifying de novo free fatty acid synthesis, and improving mitochondrial function. On the other hand, high-intensity interval training has recently been recognized as an exercise modality that demonstrated an improvement in liver stiffness (-16.8%), these benefits appear to be independent of weight loss.15 It is important to understand that the optimal exercise prescription will vary widely among patients, depending on their physical ability, personal preferences, and even their environment.

Background Arterial stiffness and endothelial dysfunction present in metabolic associated fatty liver disease (MAFLD) confer increased cardiovascular risk, which represents the leading cause of mortality in this group of patients.

Mechanisms involved in the cardiovascular complications of MAFLD have recently been found to also affect cerebral blood flow altering cerebral hemodynamics in MAFLD subjects. These alerations can be detected through transcranial Doppler, which measures the medial cerebral artery blood flow and estimates the pulsatile index (IP) and resistance (IR), markers of cerebrovascular vasoconstriction These alterations are detected by transcranial Doppler, which measures the blood flow velocity of the middle cerebral artery and estimates the pulsatility index (PI) and resistance index(RI), which are markers of cerebrovascular vasoconstriction; and the respiratory retention index (RRI), which indicates cerebrovascular autoregulation. These abnormalities are related to vascular disease in MAFLD, which plays an essential role in ischemic stroke and cognitive impairment, which explains why MAFLD patients had lower scores on cognitive function tests.

Nonetheless, there are no studies evaluating the effect of lifestyle interventions (specifically exercise) on cerebral hemodynamics in patients with MAFLD, however, it has been shown that in other pathologies that share pathophysiological similarities with NAFLD there are beneficial changes in this outcome. An example of the above is chronic heart failure and liver cirrhosis, where physical exercise attenuates the inflammatory cascade (decrease in IL6, IL8, IL12, TNFa), and decreases the activation of the renin-angiotensin system with a direct effect on endothelial function improvement. A previous report showed that a 12-week physical training program acts on this mechanism and has a beneficial effect on cerebral hemodynamics evaluated by transcranial Doppler in patients with liver cirrhosis, which leads to an improvement in neuropsychometric tests.

Therefore, improvement in the previously described pathways through a 16-week physical training program in MAFLD patients could potentially improve alterations in cerebral blood flow, cognitive function, endothelial function, body composition, and the degree of liver steatosis and fibrosis. This outcome has never been assessed in MAFLD patients undergoing exercise. In addition, although there are studies that demonstrate the impact of diet and exercise, most have evaluated these interventions individually, which represents a limitation when implementing them as a multidisciplinary intervention.

Therefore a 16-week physical training program will decrease the pulsatility index and resistance index (cerebral hemodynamics parameters) in patients with metabolic-associated fatty liver compared to the control group without a physical training program.

AIM To evaluate the effect of a 16-week physical training program on cerebral hemodynamics in patients with fatty liver disease associated with metabolic dysfunction.

Specific objectives

1. To evaluate the effect of a 16-week physical training program compared to a control group on cerebral hemodynamics assessed by transcranial Doppler in patients with MAFLD.
2. To evaluate the effect of a physical training program for 16 weeks compared to a control group on the neuropsychometric function of patients with fatty liver disease associated with metabolic dysfunction.

Secondary Objectives

1. To assess the effect of a physical training program for 16 weeks compared to a control group on endothelial function assessed by pulse rate testing in patients with MAFLD.
2. To evaluate the effect of a physical training program for 16 weeks compared to a control group on liver enzymes and the degree of liver steatosis and fibrosis evaluated by transient elastography in fatty liver disease associated with metabolic dysfunction.
3. To assess the effect of a physical training program for 16 weeks compared to a control group on the body composition of patients with MAFLD.

Methodology Population and place of study Outpatients with MAFLD from the gastroenterology service of the Salvador Zubirán National Institute of Medical Sciences and Nutrition.

Location Department of Gastroenterology, Department of Neurology and Metabolic Diseases Research Unit (UIEM), Salvador Zubirán National Institute of Medical Sciences and Nutrition.

Sample size and sampling type n= 18 per group (2)= 36 (.20) = 36 (21 per group) It is necessary to include 21 patients in each group considering a 20% loss if it is desired to obtain an 80% chance of detecting a difference in the pulsatility/resistance index of the middle cerebral artery or more between the two treatment groups.

Assignment of arms

At baseline, patients will be randomized into two groups, using the block sequence of three. The groups are:

* Control: Nutritional treatment with caloric restriction and mental exercise.
* Intervention: Nutritional treatment with caloric restriction, mental exercise, and physical training program.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with a diagnosis of MAFLD (biopsy and/or imaging and clinical context).

  * Both sexes.
  * Age 18-60 years.
  * BMI >30Kg/m2.
  * Not having participated in another intervention protocol for MAFLD in the previous three months.
  * Patients who agree to participate and sign the informed consent.

Exclusion Criteria:

* Heart failure.

  * Uncontrolled DM2, diabetic complications, known peripheral vascular disease, or neuropathy.
  * Cancer.
  * Orthopedic inability to exercise.
  * With advanced liver fibrosis (>F2), estimated by transient elastography.
  * Loss of >10% of their body weight in the last three months.
  * Consumption of supplements/food supplements and/or current or previous significant consumption of alcohol for more than three previous consecutive months (>30 g in women and >40 g in men).
  * Patients with neurological disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Chage in Pulsatility index (PI) of the middle cerebral artery | The first measurement occurs at the baseline visit and the last measurement at the sixteenth week for a total of 18 weeks between the first and last measurement.
  The pulsatility index (PI) of the middle cerebral artery is a calculated parameter in doppler ultrasound, derived from the maximum, minimum, and mean Doppler frequency shifts during a defined cardiac cycle. Along with resistive index (RI), it is typically used to assess the resistance in a pulsatile vascular system.
Change in Resistance index (RI) of the middle cerebral artery | The first measurement occurs at the baseline visit and the last measurement at the sixteenth week for a total of 18 weeks between the first and last measurement.
  RI is a calculated flow parameter in doppler ultrasound of the of the middle cerebral artery, derived from the maximum, minimum, and mean Doppler frequency shifts during a defined cardiac cycle. Along with the pulsatility index (PI), it is typically used to assess the resistance in a pulsatile vascular system.

SECONDARY OUTCOMES:
Change in Liver steatosis | The first measurement occurs at the baseline visit and the last measurement at the sixteenth week for a total of 18 weeks between the first and last measurement.
  Liver steatosis can be measure by transient elastography (FibroScan). The CAP score is a measurement of fatty change in the liver. The CAP score is measured in decibels per meter (dB/m). It ranges from 100 to 400 dB/m; using these measurements we classify fatty liver in grades.
Change in Liver fibrosis | The first measurement occurs at the baseline visit and the last measurement at the sixteenth week for a total of 18 weeks between the first and last measurement.
  The fibrosis result is measured in kilopascals (kPa).
Change in BMI (kg/m^2) | The first measurement is at the baseline visit, then at week 1, week 4, week 8, week 12, and week 16, for a total of 18 weeks between the first and last measurement
  Two nutritionists will measure the weight (kg), height (meters) to calculate BMI (kg/m^2)
Change in Endothelial function | The first measurement occurs at the baseline visit and the last measurement at the sixteenth week for a total of 18 weeks between the first and last measurement.
  The vascular endothelial function will be evaluated using the simultaneous carotid-femoral tonometry method through the pulse wave velocity (PWV) test, which represents a non-invasive measurement of arterial stiffness.
Change in Cognitive evaluation | The first measurement occurs at the baseline visit and the last measurement at the sixteenth week for a total of 18 weeks between the first and last measurement.
  The Montreal Cognitive Assessment (MoCA) will be applied, which is a cognitive assessment instrument that assesses the domains: attention and concentration; executive functions, memory, language, visuospatial skills, reasoning, calculation, and orientation.
Change in IL-1B | The first measurement is made two weeks before initiating the trial, then at week 1, week 4, week 8, week 12, and week 16, for a total of 18 weeks between the first and last measurement.
  A peripheral blood sample will be obtained at each visit, stored, and subsequently measured ( IL-1B)
Change in IL-6 | The first measurement is made two weeks before initiating the trial, then at week 1, week 4, week 8, week 12, and week 16, for a total of 18 weeks between the first and last measurement.
  A peripheral blood sample will be obtained at each visit, stored, and subsequently measured ( IL-6)
Change in TNF-a | The first measurement is made two weeks before initiating the trial, then at week 1, week 4, week 8, week 12, and week 16, for a total of 18 weeks between the first and last measurement.
  A peripheral blood sample will be obtained at each visit, stored, and subsequently measured ( TNF-a)
Change in 8-hydroxydeoxyguanosine (8-OHdG) | The first measurement is made two weeks before initiating the trial, then at week 1, week 4, week 8, week 12, and week 16, for a total of 18 weeks between the first and last measurement.
  A peripheral blood sample will be obtained at each visit, stored, and subsequently measured ( 8-hydroxydeoxyguanosine (8-OHdG))

OTHER OUTCOMES:
Change in Resting energy expenditure (REE) | Only at the baseline visit (week 1)
  Resting energy expenditure (REE) will be measured using indirect calorimetry.
Change in number of steps/day | The first measurement is made two weeks before initiating the trial, then at week 1, week 4, week 8, week 12, and week 16, for a total of 18 weeks between the first and last measurement.
  At the baseline visit, a count will be made of the average number of steps that the subjects took in a period of two previous weeks. This activity will be supervised through the polar loop pedometer bracelet that patients will have to wear throughout the protocol.
change in microbiota diversity. | The first measurement is made two weeks before initiating the trial and at week 16, for a total of 18 weeks between the first and last measurement
  Diversity of microbiota will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Macías-Rodríguez, MD,MSc,PhD, Principal Investigator — Department of Gastroenterology, INCMNSZ
Locations (1):
- Instituto nacional de ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

REFERENCES:
- [Derived] Roman-Calleja BM, Ruiz-Margain A, Duarte-Rojo A, Flores-Silva F, Martinez-Cabrera CF, Gutierrez-Rosas LE, Valencia-Pena BA, Cantu-Brito C, Chalasani N, Aguilar-Salinas CA, Macias-Rodriguez RU. Physical exercise improves neurocognition in patients with metabolic dysfunction-associated steatotic liver disease. Liver Transpl. 2025 Nov 3. doi: 10.1097/LVT.0000000000000767. Online ahead of print. PMID 41182078